CLINICAL TRIAL: NCT07116967
Title: A Phase 3b/4 Multi-center, Randomized, Open-label, Long-term Safety Study of Deucravacitinib in Comparison to Ustekinumab in Participants With Moderate-to-Severe Plaque Psoriasis
Brief Title: Long-Term Safety Study of Deucravacitinib Versus Ustekinumab in Participants With Psoriasis (PRAGMATYK)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IM011-1130; U1111-1291-5815 (Other: WHO); 2023-503766-24 (Other: EU CTR)
Record Dates: First submitted 2025-08-04; First posted 2025-08-12 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Plaque Psoriasis
Keywords: Deucravacitinib; Plaque psoriasis; Cardiovascular risk; PRAGMATYK
MeSH Terms: interventions — deucravacitinib; Ustekinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental)
  Interventions: Drug: Deucravacitinib
- Arm B (Active Comparator)
  Interventions: Drug: Ustekinumab

INTERVENTIONS:
Drug: Deucravacitinib — Specified dose on specified days
  Other Names: SOTYKTU
  Arms: Arm A
Drug: Ustekinumab — Specified dose on specified days
  Arms: Arm B

SUMMARY:
A study to evaluate the long-term safety of Deucravacitinib versus Ustekinumab in participants with psoriasis

ELIGIBILITY:
Inclusion Criteria:

* Participants with moderate-to-severe plaque psoriasis:

  1. Deemed by the Investigator to be a candidate for phototherapy or systemic treatment for psoriasis, including ustekinumab;
  2. Have at least 1 of the following cardiovascular risk factors:
* Current cigarette smoker
* Diagnosis of hypertension
* Diagnosis of hyperlipidemia
* Diabetes mellitus type 1 or 2
* History of one or more of the following cardiovascular events: Coronary intervention (PCI) or coronary artery bypass grafting (CABG), myocardial infarction (heart attack), cardiac arrest, hospitalization for unstable angina, acute coronary syndrome, stroke, or transient ischemic attack
* Obesity
* Family history of premature coronary heart disease or sudden death in a first-degree male relative younger than 55 years of age or in a first-degree female relative younger than 65 years of age.

Exclusion Criteria:

* Participants must not have recent history of 1 of the following cardiovascular events: MI, stroke, or coronary revascularization, or VTE within 90 days prior to Day 1.
* Participants must not have unstable CVD, defined as a recent clinical cardiovascular event (eg, unstable angina, rapid atrial fibrillation), or a cardiac hospitalization (eg, pacemaker implantation, HF) within 90 days prior to Day 1.
* Participants must not have evidence of active cancer or history of cancer (solid organ or hematologic malignancy including myelodysplastic syndrome) or lymphoproliferative disease within the previous 5 years (other than resected cutaneous basal cell or squamous cell carcinoma, or carcinoma of cervix in situ that has been treated with no evidence of recurrence).
* Other protocol define inclusion/exclusion criteria apply.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3040 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2031-01-16 (Estimated); Study Completion 2031-01-16 (Estimated)

PRIMARY OUTCOMES:
Composite cardiovascular adjudicated 3-point major adverse cardiovascular event (MACE) plus coronary revascularization | Up to 5 years
  MACE defined as non-fatal myocardial infarction [MI], nonfatal stroke, and cardiovascular death

SECONDARY OUTCOMES:
Number of participants with non-fatal MI | Up to 5 years
Number of participants with non-fatal stroke | Up to 5 years
Death due to cardiovascular events | Up to 5 years
Number of participants with coronary revascularization | Up to 5 years
Number of participants with 3-point MACE (non-fatal MI, non-fatal stroke, and cardiovascular death) | Up to 5 years
Number of participants with pulmonary embolism (PE) | Up to 5 years
Number of participants with deep vein thrombosis (DVT) | Up to 5 years
Number of participants with composite venous thromboembolism (VTE) | Up to 5 years
  PE, DVT and retinal vein occlusion
Number of participants with arterial thromboembolic events (including retinal artery occlusion) | Up to 5 years
Number of participants with heart failure (HF) requiring hospitalization or urgent visit | Up to 5 years
Number of participants with Malignancy excluding non-melanoma skin cancer (NMSC) | Up to 5 years
Number of participants with NMSC | Up to 5 years
Number of participants with opportunistic infections | Up to 5 years
  Opportunistic infections include tuberculosis and complicated herpes zoster (eg, disseminated herpes zoster, affecting more than 2 dermatomes, ophthalmic or meningoencephalopathic involvement, and other atypical presentations)
Number of participants with Serious AEs (SAEs) | Up to 60 days after last dose
All-cause mortality | Up to 60 days after last dose
AEs leading to permanent treatment discontinuation | Up to 60 days after last dose
Change from baseline in liver function test | Up to 60 days after last dose
Change from baseline in fasting lipid panel | Up to 60 days after last dose

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (332):
- United States (108):
  - Local Institution - 0088, Birmingham, Alabama
  - Medical Dermatology Specialists - Phoenix, Phoenix, Arizona
  - Local Institution - 0495, Phoenix, Arizona
  - Omni Dermatology, Phoenix, Arizona
  - Alliance Dermatology, Phoenix, Arizona
  - Local Institution - 0322, Scottsdale, Arizona
  - Local Institution - 0188, Scottsdale, Arizona
  - Scottsdale Clinical Trials, Scottsdale, Arizona
  - Omni Dermatology, Tempe, Arizona
  - Clinical Trials Institute of Northwest Arkansas, Fayetteville, Arkansas
  - T. Joseph Raoof MD Inc, Encino, California
  - Center For Dermatology Clinical Research, Inc., Fremont, California
  - Marvel Clinical Research, Huntington Beach, California
  - Dermatology Research Associates - Howard Sofen, MD, Los Angeles, California
  - Local Institution - 0192, Los Angeles, California
  - Northridge Clinical Trials - Elite Clinical Network, Northridge, California
  - Cura Clinical Research - Palmdale, Palmdale, California
  - Pasadena Clinical Trials, Pasadena, California
  - Empire Clinical Research - Pomona, Pomona, California
  - Local Institution - 0316, Sacramento, California
  - Local Institution - 0038, Sacramento, California
  - Local Institution - 0078, San Diego, California
  - Cura Clinical Research - Santa Clarita, Santa Clarita, California
  - Clinical Science Institute, Santa Monica, California
  - Advanced Dermatology and Skin Cancer Institute - Beverly Hills, Sherman Oaks, California
  - Unison Clinical Trials, Sherman Oaks, California
  - Local Institution - 0181, Walnut Creek, California
  - Local Institution - 0494, Castle Rock, Colorado
  - Local Institution - 0334, Washington D.C., District of Columbia
  - Skin Care Research LLC (SCR) - Boca Raton, Boca Raton, Florida
  - Driven Research LLC, Coral Gables, Florida
  - Florida Academic Dermatology Center, Coral Gables, Florida
  - Accel Research Sites - Maitland Clinical Research Unit, Maitland, Florida
  - Miami Dermatology and Laser Research, Miami, Florida
  - International GCC Research, Miami, Florida
  - Local Institution - 0493, Miami, Florida
  - Local Institution - 0029, Miami Lakes, Florida
  - Renstar Medical Research, Ocala, Florida
  - LENUS Research, Sweetwater, Florida
  - Local Institution - 0089, Tampa, Florida
  - Dermatology Affiliates Research Institute, Atlanta, Georgia
  - Local Institution - 0419, Savannah, Georgia
  - Local Institution - 0395, Chicago, Illinois
  - Endeavor Health Clinical Trials, Skokie, Illinois
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - Southern Indiana Clinical trials, New Albany, Indiana
  - Equity Medical - Bowling Green, Bowling Green, Kentucky
  - Local Institution - 0030, Owensboro, Kentucky
  - Clinical Trials Management, LLC - Northshore Office, Covington, Louisiana
  - Shondra L. Smith, MD - Dermatology and Advanced Aesthetics, Lake Charles, Louisiana
  - Clinical Trials Management, Metairie, Louisiana
  - Local Institution - 0069, New Orleans, Louisiana
  - Local Institution - 0331, Rockville, Maryland
  - Metro Boston Clinical Partners, Brighton, Massachusetts
  - Kuchnir Dermatology & Dermatologic Surgery, Milford, Massachusetts
  - Local Institution - 0287, Quincy, Massachusetts
  - Michigan Center for Skin Care Research, Clinton Township, Michigan
  - Somerset Skin Centre, Troy, Michigan
  - Minnesota Clinical Study Center (MCSC), New Brighton, Minnesota
  - Local Institution - 0433, Columbia, Missouri
  - Local Institution - 0397, Omaha, Nebraska
  - Local Institution - 0454, Las Vegas, Nevada
  - Las Vegas Clinical Trials, LLC, North Las Vegas, Nevada
  - Local Institution - 0097, Portsmouth, New Hampshire
  - StracSkin, Portsmouth, New Hampshire
  - Local Institution - 0079, Teaneck, New Jersey
  - Schweiger Dermatology, Verona, New Jersey
  - Forest Hills Dermatology Group, Kew Gardens, New York
  - The Skin Center Dermatology Group, New City, New York
  - Local Institution - 0410, New York, New York
  - Skin Search Rochester, Rochester, New York
  - Equity Medical - New York, The Bronx, New York
  - Accellacare - Cary, Cary, North Carolina
  - Local Institution - 0332, Chapel Hill, North Carolina
  - Local Institution - 0165, Chapel Hill, North Carolina
  - Hickory Dermatology Research Center, Hickory, North Carolina
  - Wilmington Dermatology Center-WDC Cosmetic and Research, Wilmington, North Carolina
  - Local Institution - 0177, Bexley, Ohio
  - Local Institution - 0392, Canal Winchester, Ohio
  - Apex Clinical Research Center - Canton, Canton, Ohio
  - Local Institution - 0182, Fairborn, Ohio
  - Apex Clinical Research Center, Mayfield Heights, Ohio
  - Local Institution - 0436, Medina, Ohio
  - Unity Clinical Research (UCR), Oklahoma City, Oklahoma
  - Velocity Clinical Research, Medford, Medford, Oregon
  - Local Institution - 0180, Portland, Oregon
  - Oregon Dermatology and Research Center, Portland, Oregon
  - Best Skin Research, Camp Hill, Pennsylvania
  - Local Institution - 0131, Exton, Pennsylvania
  - UPMC Department of Dermatology, Pittsburgh, Pennsylvania
  - Palmetto Clinical Trial Services - Administrative Office, Anderson, South Carolina
  - Local Institution - 0422, Greenville, South Carolina
  - Palmetto Clinical Trial Services - Administrative Office, Greenville, South Carolina
  - Local Institution - 0418, North Charleston, South Carolina
  - Local Institution - 0084, Rapid City, South Dakota
  - Discover Dermatology, LLC d/b/a Goodlettsville Dermatology Research, Goodlettsville, Tennessee
  - Cumberland Skin Center for Clinical Research, Hermitage, Tennessee
  - International Clinical Research (IC Research) - Murfreesboro, Murfreesboro, Tennessee
  - Belle Meade Dermatology Research, Nashville, Tennessee
  - Arlington Center for Dermatology, Arlington, Texas
  - Studies in Dermatology, LLC, Cypress, Texas
  - Modern Research Associates, PLLC, Dallas, Texas
  - Local Institution - 0468, Dallas, Texas
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
  - Center For Clinical Studies, Webster, Texas
  - Local Institution - 0333, Norfolk, Virginia
  - Frontier Dermatology, Mill Creek, Washington
  - Premier Clinical Research, Spokane, Washington
- Argentina (12):
  - Consultorios Reumatológicos Pampa, C.a.b.a., Buenos Aires
  - Local Institution - 0429, Buenos Aires, Buenos Aires F.D.
  - Instituto de Neumonologia y Dermatologia, Buenos Aires, Buenos Aires F.D.
  - Buenos Aires Skin S.A, Buenos Aires, C
  - STAT Research S.A., Ciudad Autonoma Buenos Aires, C
  - Psoriahue, Ciudad Autonoma Buenos Aires, C
  - CEMEDIAB - Centro Medico Diabetologico, Ciudad Autónoma Buenos Aires, C
  - Derma Internacional S.A., Autonomous City of Buenos Aires
  - CONEXA Investigacion Clinica S.A., Buenos Aires
  - Local Institution - 0474, Buenos Aires
  - Instituto de Investigaciones Clínicas Córdoba S.A., Córdoba
  - Viviana Parra Instituto Parra Dermatología, Mendoza
- Australia (8):
  - The Skin Hospital, Darlinghurst, New South Wales
  - St George Dermatology & Skin Cancer Centre, Kogarah, New South Wales
  - Local Institution - 0216, Westmead, New South Wales
  - Local Institution - 0285, Woolloongabba, Queensland
  - Local Institution - 0311, Woolloongabba, Queensland
  - Skin Health Institute Inc., Carlton, Victoria
  - Local Institution - 0345, Clayton, Victoria
  - Dr Rodney Sinclair Pty Ltd., East Melbourne, Victoria
- Belgium (3):
  - Local Institution - 0063, Woluwe-Saint-Lambert, BRU
  - Local Institution - 0243, Maldegem, Oost- Vlaanderen
  - Local Institution - 0239, Ghent, VOV
- Brazil (13):
  - Local Institution - 0037, Juiz de Fora, Minas Gerais
  - Local Institution - 0416, Curitiba, Paraná
  - Local Institution - 0384, Curitiba, Paraná
  - Local Institution - 0385, João Pessoa, Paraíba
  - Local Institution - 0390, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0036, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0399, Botucatu, São Paulo
  - Local Institution - 0383, Campinas, São Paulo
  - Local Institution - 0193, Ribeirão Preto, São Paulo
  - Local Institution - 0400, São José do Rio Preto, São Paulo
  - Local Institution - 0490, Vila Clementino, São Paulo-SP
  - Local Institution - 0039, São Paulo
  - Local Institution - 0450, São Paulo
- Bulgaria (9):
  - Local Institution - 0481, Burgas
  - Local Institution - 0480, Lovech
  - Local Institution - 0479, Pleven
  - Local Institution - 0483, Plovdiv
  - Local Institution - 0486, Plovdiv
  - Local Institution - 0482, Rousse
  - Local Institution - 0487, Sofia
  - Local Institution - 0484, Sofia
  - Local Institution - 0485, Stara Zagora
- Canada (32):
  - Local Institution - 0013, Calgary, Alberta
  - Local Institution - 0126, Calgary, Alberta
  - Beacon Dermatology, Calgary, Alberta
  - Stratica Dermatology, Edmonton, Alberta
  - Alberta Dermasurgery Centre, Edmonton, Alberta
  - Vida Clinic Research, Edmonton, Alberta
  - Interior Dermatology Centre, Kelowna, British Columbia
  - Skin Care West, Nanaimo, British Columbia
  - Local Institution - 0120, Surrey, British Columbia
  - Enverus Medical Research, Surrey, British Columbia
  - Wiseman Dermatology Research Inc., Winnipeg, Manitoba
  - Dr Tracey Brown-Maher Dermatology Clinic and Research Centre, St. John's, Newfoundland and Labrador
  - CCA Medical Research, Ajax, Ontario
  - SimcoDerm Medical and Surgical Dermatology Center, Barrie, Ontario
  - Local Institution - 0005, Hamilton, Ontario
  - Centricity Research London Victoria Multispecialty, London, Ontario
  - Lovegrove Dermatology, London, Ontario
  - DermEffects, London, Ontario
  - Lynderm Research Inc., Markham, Ontario
  - DermEdge, Mississauga, Ontario
  - Ryan Clinical Research Inc, Newmarket, Ontario
  - North Bay Dermatology Centre, North Bay, Ontario
  - The Centre for Clinical Trials Inc., Oakville, Ontario
  - Local Institution - 0003, Ottawa, Ontario
  - SKiN Centre for Dermatology, Peterborough, Ontario
  - The Centre for Dermatology, Richmond Hill, Ontario
  - North York Research Inc., Toronto, Ontario
  - Toronto Research Centre, Toronto, Ontario
  - Centre de Recherche Saint-Louis, Montreal, Quebec
  - Centre de Recherche Saint-Louis, Sherbrooke, Quebec
  - Sima Recherche, Verdun, Quebec
  - Centre de Recherche Saint-Louis, Québec
- Chile (4):
  - Local Institution - 0463, Viña del Mar, Reñaca Norte
  - Local Institution - 0462, Santiago, Santiago Metropolitan
  - Local Institution - 0461, Santiago, Santiago Metropolitan
  - Local Institution - 0459, Santiago, Santiago Metropolitan
- China (28):
  - Local Institution - 0352, Bengbu, Anhui
  - Local Institution - 0050, Beijing, Beijing Municipality
  - Local Institution - 0140, Beijing, Beijing Municipality
  - Local Institution - 0226, Chongqing, Chongqing Municipality
  - Local Institution - 0049, Fuzhou, FJ
  - Local Institution - 0353, Guangzhou, Guangdong
  - Local Institution - 0129, Shenzhen, Guangdong
  - Local Institution - 0438, Shijiazhuang, Hebei
  - Local Institution - 0293, Harbin, Heilongjiang
  - Local Institution - 0439, Zhengzhou, Henan
  - Local Institution - 0047, Wuhan, Hubei
  - Local Institution - 0046, Wuhan, Hubei
  - Local Institution - 0414, Wuhan, Hubei
  - Local Institution - 0356, Zhenjiang, Jiangsu
  - Local Institution - 0417, Changchun, Jilin
  - Local Institution - 0054, Shenyang, Liaoning
  - Local Institution - 0055, Taiyuan, Shan1xi
  - Local Institution - 0194, Jinan, Shandong
  - Local Institution - 0108, Jinan, Shandong
  - Local Institution - 0354, Chengdu, Sichuan
  - Local Institution - 0053, Chengdu, Sichuan Provience
  - Local Institution - 0044, Hangzhou, Zhejiang
  - Local Institution - 0277, Hangzhou, Zhejiang
  - Local Institution - 0052, Ningbo, Zhejiang
  - Local Institution - 0207, Changsha Shi
  - Local Institution - 0051, Hangzhou
  - Local Institution - 0401, Nanjing
  - Local Institution - 0386, Shenzhen
- Czechia (6):
  - Local Institution - 0202, Prague, PR
  - Local Institution - 0440, Brno
  - Local Institution - 0151, Olomouc
  - Local Institution - 0389, Prague
  - Local Institution - 0121, Prague
  - Local Institution - 0150, Ústí nad Labem
- Denmark (4):
  - Local Institution - 0196, Copenhagen, Capital Region
  - Local Institution - 0324, Aarhus
  - Local Institution - 0290, Hellerup
  - Local Institution - 0457, Herlev
- France (3):
  - Local Institution - 0238, Nantes
  - Local Institution - 0153, Nice
  - Local Institution - 0217, Rennes
- Germany (23):
  - Local Institution - 0101, Freiburg im Breisgau, Baden-Wurttemberg
  - Local Institution - 0127, Langenau, Baden-Wurttemberg
  - Local Institution - 0299, Mahlow, Brandenburg
  - Local Institution - 0117, Witten, Northwest
  - Local Institution - 0237, Mainz, Rhineland-Palatinate
  - Local Institution - 0245, Quedlinburg, Saint
  - Local Institution - 0255, Dresden, Saxony
  - Local Institution - 0382, Leipzig, Saxony
  - Local Institution - 0340, Kiel, Schleswig-Holstein
  - Local Institution - 0291, Berlin, State of Berlin
  - Local Institution - 0476, Berlin
  - Local Institution - 0001, Bramsche
  - Local Institution - 0109, Dresden
  - Local Institution - 0200, Erlangen
  - Local Institution - 0130, Frankfurt am Main
  - Local Institution - 0473, Friedrichshafen
  - Local Institution - 0472, Halle
  - Local Institution - 0471, Hamburg
  - Local Institution - 0106, Heidelberg
  - Local Institution - 0115, Mainz
  - Local Institution - 0112, Memmingen
  - Local Institution - 0295, Merzig
  - Local Institution - 0260, Tübingen
- Hungary (4):
  - Local Institution - 0206, Szeged, Csongrád megye
  - Local Institution - 0209, Budapest
  - Local Institution - 0266, Debrecen
  - Local Institution - 0404, Veszprém
- Italy (5):
  - Local Institution - 0269, L’Aquila, AQ
  - Local Institution - 0305, Modena, MO
  - Local Institution - 0307, Bologna
  - Local Institution - 0249, Naples
  - Local Institution - 0309, Roma
- Japan (14):
  - Nagoya City University Hospital, Nagoya-sh, Aichi-ken
  - Local Institution - 0451, Toyoake Shi, Aichi-ken
  - Local Institution - 0374, Asahikawa-shi, Hokkaido
  - Local Institution - 0378, Suita, Osaka
  - Local Institution - 0377, Suita-shi, Osaka
  - Local Institution - 0452, Ōtsu, Shiga
  - St. Luke's International Hospital, Chūōku, Tokyo-to
  - Local Institution - 0376, Gifu
  - Local Institution - 0391, Itabashi-Ku
  - Local Institution - 0375, Kanazawa
  - Local Institution - 0379, Kurume, Fukuoka
  - Local Institution - 0456, Okayama
  - Local Institution - 0380, Sakaishi
  - Local Institution - 0415, Sakaishi
- Mexico (8):
  - Local Institution - 0467, Mexicali, Estado de Baja California
  - Local Institution - 0321, Guadalajara, Jalisco
  - Local Institution - 0470, Zapopan, Jalisco
  - Local Institution - 0113, Monterrey, Nuevo León
  - Local Institution - 0469, Monterrey, Nuevo León
  - Local Institution - 0118, Mérida, Yucatán
  - Local Institution - 0466, Chihuahua City
  - Local Institution - 0465, Mexico City
- Poland (19):
  - Local Institution - 0265, Torun, Kuyavian-Pomeranian Voivodeship
  - Local Institution - 0425, Puławy, Lublin Voivodeship
  - Local Institution - 0424, Warsaw, Masovian Voivodeship
  - Local Institution - 0252, Rzeszów, Podkarpackie Voivodeship
  - Local Institution - 0292, Bialystok, Podlaskie Voivodeship
  - Local Institution - 0195, Katowice, Silesian Voivodeship
  - Local Institution - 0423, Olsztyn, Warmian-Masurian Voivodeship
  - Local Institution - 0428, Poznan, Wielkopolska
  - Local Institution - 0296, Bialystok
  - Local Institution - 0091, Gdansk
  - Local Institution - 0444, Gdynia
  - Local Institution - 0162, Katowice
  - Local Institution - 0154, Katowice
  - Local Institution - 0276, Lodz
  - Local Institution - 0413, Mikołów
  - Local Institution - 0421, Skierniewice
  - Local Institution - 0308, Warsaw
  - Local Institution - 0205, Wroclaw
  - Local Institution - 0244, Kielce, Świętokrzyskie Voivodeship
- Centro Reumatologico Caguas, Caguas, Puerto Rico
- Romania (9):
  - Local Institution - 0405, Craiova, Dolj
  - Local Institution - 0403, Iași, IS
  - Local Institution - 0388, Reghin, MS
  - Local Institution - 0441, Timișoara, Timiș County
  - Local Institution - 0225, Brasov
  - Local Institution - 0412, Bucharest
  - Local Institution - 0402, Bucharest
  - Local Institution - 0398, Constanța
  - Local Institution - 0458, Iași
- South Korea (3):
  - Local Institution - 0065, Seongnam-si, Gyeonggi-do, Gyeonggi-do
  - Local Institution - 0067, Seongnam-si
  - Local Institution - 0060, Seoul
- Spain (5):
  - Local Institution - 0337, Las Palmas de Gran Canaria, Las Palmas
  - Local Institution - 0242, Alcorcón, Madrid
  - Local Institution - 0445, Málaga, MA
  - Local Institution - 0236, Seville, SE
  - Local Institution - 0258, Madrid
- Sweden (2):
  - Local Institution - 0211, Lund, M
  - Local Institution - 0223, Borås
- Taiwan (2):
  - Local Institution - 0315, Zuoying Dist, Kaohsiung
  - National Taiwan University Hospital, Taipei
- United Kingdom (7):
  - Velocity Clinical Research, High Wycombe, High Wycombe, Bucks
  - Local Institution - 0284, Dunfermline, FIF
  - Velocity Clinical Research - North London, London, Greater London
  - University Hospital Southampton NHS Foundation Trust - Southampton General Hospital, Southampton, Hampshire
  - Local Institution - 0241, London, LND
  - Salford Care Organisation, Salford, SLF
  - Local Institution - 0499, Bristol, South West

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT07116967.html